CLINICAL TRIAL: NCT00591682
Title: Phase I Dose Escalation Study to Determine the Safety and Pharmacokinetics of MSX-122 Administered Orally in Patients With Refractory Metastatic or Locally Advanced Solid Tumors
Brief Title: MSX-122 Administered Orally in Patients With Refractory Metastatic or Locally Advanced Solid Tumors
Status: Suspended | Phase: Phase 1 | Type: Interventional
Sponsor: Metastatix, Inc. (Industry)
Responsible Party: Carol G. Gallagher, Pharm. D., Metastatix, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0407
Record Dates: First submitted 2007-12-31; First posted 2008-01-11 (Estimated); Last update posted 2008-03-26 (Estimated); Status verified 2008-03

CONDITIONS: Solid Tumors
MeSH Terms: interventions — N,N'-(1,4-phenylenebis(methylene))dipyrimidin-2-amine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): MSX-122
  Interventions: Drug: MSX-122

INTERVENTIONS:
Drug: MSX-122 — Dosage form = capsule
  Starting Dose (First Patient Cohort - Dose Level 1) = 50 mg taken orally once daily, 7 days per week for 4 weeks (total of 28 days), followed immediately by a second course of 28 days with identical dosage form and schedule. (Each patient in each cohort treated for a minimum of 56 days, unless obviated by toxicity.)
  * If there is no evidence of toxicity at the current dose level, then the dose of MSX-122 will be increased by 100% for the next patient cohort.
  * If a grade 1-2 toxicity is observed, then the dose will be increased by 50% for the next patient cohort.
  * If a grade 3 toxicity (non-dose limiting toxicity) is observed then the dose will be increased by 25% for the next patient cohort.

SUMMARY:
Primary Objectives:

1. To determine the maximum tolerated dose (MTD) and the recommended Phase II dose(s) and schedule of MSX-122
2. To characterize the dose limiting toxicities (DLTs) and determine the overall safety and tolerability of MSX-122

Secondary Objectives:

1. To determine the pharmacokinetics and pharmacodynamics of orally administered MSX-122
2. To evaluate the preliminary evidence for anti-tumor activity of MSX-122
3. To perform correlative studies to elucidate signaling pathways involved in CXCR4 activation in blood and optional tissue specimens by IHC (immunohistochemistry) and RPPA (reverse phase protein microarrays)

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically confirmed advanced malignancy that is metastatic or unresectable and which is refractory to standard therapy or for which there is no standard therapy that provides benefit
* Measurable or non-measurable disease at baseline
* At least four weeks since the last dose of prior chemotherapy, treatment with biologic agents, radiation therapy or investigational agents
* Patients must have recovered from the adverse effects of prior therapy at the time of enrollment to a grade one or less(excluding alopecia)
* Patient will not be treated with any other chemotherapy, immunotherapy, radiotherapy or investigational drug while enrolled on this protocol
* Age >/= 18 year, male or female patients
* Eastern Cooperative Oncology Group (ECOG) performance status 0,1, or 2
* Life expectancy of greater than 3 months following study entry
* Adequate renal function, defined by serum creatinine less than or equal to 1.5 x ULN
* Adequate hepatic function as defined by aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels </= to 2.5 x ULN and total bilirubin </= to 1.5 x ULN. In the presence of liver metastasis, adequate hepatic function is defined as ALT and AST </= 5 x ULN and total bilirubin </= 3 x ULN. Alkaline phosphatase levels less than or equal to 2.5 x ULN. In the presence of extensive bone metastases, alkaline phosphatase is defined as less than or equal to 5 x ULN
* Adequate bone marrow function as defined by an absolute neutrophil count of >/= 1,500/mm3 (>/=1.5 x 10^9/L), platelet count of >/= 100,000/mm3 (>/=100 x10^9/L) and hemoglobin of >/= 8 gm/dL
* Left ventricular ejection fraction of 50% or greater as measured by echocardiogram or MUGA
* For women of childbearing potential, a negative serum pregnancy test result at screening
* Women of child-bearing potential or men whose sexual partners are women of child-bearing potential must agree to use two methods of adequate contraception (e.g. hormonal and barrier method of birth control) prior to study entry, for the duration of the study, and for 21 days after the last dose of study medication. Acceptable methods of contraception include condoms, diaphragm ,birth control pills, birth control patch, hormonal injections, intrauterine device (IUD), surgical sterilization and/or under the skin implants
* Signed and dated institutional review board (IRB)-approved informed consent before any protocol-specific screening procedures are performed

Exclusion Criteria:

* Patients with uncontrolled concurrent illness, including but not limited to: ongoing or active infection; uncontrolled arterial hypertension (>/= 140/90 mm of mercury on medications); uncontrolled endocrine diseases (e.g. diabetes mellitus, hypothyroidism or hyperthyroidism, adrenal disorder); altered mental status or psychiatric illness/social situations that would limit compliance with study requirements and/or obscure study results
* Patients with a history of a cardiovascular illness including but not confined to: CHF (grade III or IV NYHA); a history of angina pectoris within the previous year; history of any cardiac arrhythmia; QTc prolongation as determined by Bazett's formula and defined as QTc interval >480 msec (including patients on medication which may prolong QTc), or history of myocardial infarction within one year of study enrollment
* Patients with leukemias or myelodysplastic syndrome (MDS)
* Immunocompromised patients, including subjects known to be infected by human immunodeficiency virus (HIV)
* Patients with a history of autologous BMT within the previous five years. Patients with organ transplants, or allogeneic BMT will not be eligible for the study
* Patients with untreated or uncontrolled brain metastasis, or patients with leptomeningeal disease
* Patients unable to swallow oral medications or with pre-existing gastrointestinal disorders that might interfere with proper absorption of the oral drugs (e.g. WDHA syndrome, carcinoid syndromes, diarrhea due to infections, malabsorption syndromes secondary to surgery or chemotherapy).
* Patients with a history of major surgery within 28 days of first receipt of study drug
* Nursing or pregnant women
* Patients with any other diseases, metabolic dysfunction, physical examination finding or clinical laboratory finding that in the opinion of the investigator, contraindicates the use of an investigational drug, or that may render the patient at excessively high risk for treatment complications
* Patients with a history of one or more other primary carcinomas
* Patients with a known hypersensitivity to any of the components of the drug product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2007-11; Primary Completion 2008-12 (Estimated); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose (MTD) and the recommended Phase II dose(s) and schedule of MSX-122 | 12 Months Estimated
Characterize the dose limiting toxicities (DLTs) and determine the overall safety and tolerability of MSX-122 | 12 Months Estimated

SECONDARY OUTCOMES:
Determine the pharmacokinetics and pharmacodynamics of orally administered MSX-122 | 12 Months Estimated
Evaluate the preliminary evidence for anti-tumor activity of MSX-122 | 12 Months Estimated
Perform correlative studies to elucidate signaling pathways involved in CXCR4 activation in blood and optional tissue specimens by IHC (immunohistochemistry) and RPPA (reverse phase protein microarrays) | 12 Months Estimated

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer J. Wheler, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States